CLINICAL TRIAL: NCT06081205
Title: A Prospective Observational Study of Patients Admitted to a Cardiac Intensive Care Unit Due to Acute CardioVascular Disease.
Brief Title: Study of Patients Admitted to a Cardiac Intensive Care Unit With Acute CardioVascular Disease
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Katerina Naka, Professor of Cardiology, University Hospital, Ioannina
Other Study IDs: 10/270423
Record Dates: First submitted 2023-07-10; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiogenic Shock; Acute Decompensated Heart Failure; Acute Pulmonary Embolism; Acute Myocardial Infarction
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Admission in the Cardiac Intensive Care Unit (CICU) — all patients admitted in the CICU will be enrolled in the study provided they give their informed consent.
  Other Names: no further interventions

SUMMARY:
This is a registry of the patients that are admitted to CICU and treated by the Scientific Staff of the 2nd Department of Cardiology, due to an acute cardiovascular disease (acute coronary syndrome, acute heart failure, arrhythmia, pulmonary embolism, cardiac tamponade etc) in order to investigate the clinical characteristics of the patients, their outcome, identify the factors that could predict the in-hospital mortality and compare the results with the predicted by established risk scores. Furthermore, the study will investigate the one-year mortality and also the major adverse cardiac events (MACE - acute myocardial infarction, stroke, or cardiovascular death) will be measured.

DETAILED DESCRIPTION:
For every patient that will be enrolled to the study, information from the medical record will be collected, as long as he/she has provided a signed consent form after being fully informed of the study and its objectives. In case the patient cannot decide on his/her own, e.g. intubated patients, an informed consent form must be acquired by a relative or legal representative. Only the data that will be considered necessary for scientific reasons will be acquired: general and demographic information, medical information like the personal and family history, the diagnostic tests performed and the treatments or interventions that took place. The patients will not have to do anything further or undergo any additional visits or medical exams apart from those indicated; they will not receive any extra treatment (because of their participation to the study) beyond what they would receive for their condition according to the established practice so far. Furthermore, the doctor will not change or withdraw any treatment that the patients would normally receive. The patients' medical care will continue normally under the CICU doctors' supervision.

The participants will be monitored during their hospitalization in the CICU, during their hospitalization in the 2nd Department of Cardiology of the UHI after their discharge from CICU, as well as for the next 1-year in the Outpatients Clinic; if the latter is not feasible (in case of disability or distance) they will be contacted through telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Cardiac Intensive Care Unit (CICU) through the Emergency Department of the UHI
* All patients transferred to the CICU from other hospital departments or other regional secondary hospitals
* Patients with an acute cardiovascular disease that requires treatment in a CICU
* Patients who are under scientific supervision of the 2nd Department of Cardiology
* Patients (or their relative/legal representatives) that have signed the informed consent form

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that are admitted through the Emergency Department of the UHI, transferred by other hospital clinics or by other regional secondary hospitals, with an acute cardiovascular disease that requires treatment in a CICU and are under scientific supervision of the 2nd Department of Cardiology, irrespectively of gender and age. In order to be enrolled, patients or their relative/legal representative (in cases stated above) must have signed an informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2027-04-26 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | During the index admission (up to 8 weeks)
  In-hospital all-cause mortality of patients with acute cardiovascular disease that require treatment in a CICU
30-day mortality | 30 days after discharge from hospital
  30-day all-cause mortality of patients with acute cardiovascular disease that require treatment in a CICU
1-year mortality | 1-year after discharge from hospital
  1-year all-cause mortality of patients with acute cardiovascular disease that require treatment in a CICU

SECONDARY OUTCOMES:
In-hospital major adverse cardiac events (MACE) | During the index admission (up to 8 weeks)
  In-hospital MACE of patients with acute cardiovascular disease that require treatment in a CICU
30-day major adverse cardiac events (MACE) | 30 days after discharge from hospital
  30-day MACE of patients with acute cardiovascular disease that require treatment in a CICU
1-year major adverse cardiac events (MACE) | 1-year after discharge from hospital
  1-year MACE of patients with acute cardiovascular disease that require treatment in a CICU

CONTACTS AND LOCATIONS:
Overall Officials: Lampros K Michalis, MD, PhD, Study Director — Professor of Cardiology, Director of the 2nd Cardiology Department, University Hospital of Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided